CLINICAL TRIAL: NCT06866275
Title: Suramin for the Treatment of Autism Trial (STAT): A Randomized, Double Blind, Crossover Trial of KZ101 in a Male Pediatric Population With Autism Spectrum Disorder
Brief Title: Suramin for the Treatment of Autism Trial: KZ101 in a Male Pediatric Population With Autism Spectrum Disorder (ASD)
Acronym: STAT-2A
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Collaborators: Kuzani Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHOC IRB# 2308114
Record Dates: First submitted 2025-02-24; First posted 2025-03-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Suramin; suramin sodium
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Suramin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug followed by Placebo (Experimental)
  Interventions: Drug: KZ101; Drug: Placebo
- Placebo followed by Drug (Placebo Comparator)
  Interventions: Drug: KZ101; Drug: Placebo

INTERVENTIONS:
Drug: KZ101 — For active treatment with KZ101, a loading dose of 454 mg/m2 (salt-free) will be followed by a treatment dose of 363 mg/m2 (salt-free).
  Other Names: Suramin; Suramin sodium
Drug: Placebo — Dosing in the placebo group will consist of a volume of normal saline equivalent to that given during the active treatment period for each participant.
  Other Names: Saline

SUMMARY:
Suramin has been found to correct the symptoms, metabolism, and brain synaptic abnormalities in two classical genetic and environmental mouse models of autism. A preliminary clinical trial (SAT-1) examined the safety and activity of a single low-dose of suramin in children with ASD and concluded suramin showed promise as a novel approach to treatment of ASD. The current study, STAT-2A, will be a randomized, double-blind, crossover, 30-week study to evaluate the preliminary proof of concept, safety, and PK of suramin sodium (KZ101) with repeat dosing by IV infusion in males 5-14 years of age who have been diagnosed with ASD. The study will be conducted at approximately 3 sites contributing approximately 15 subjects per site. Total enrollment of approximately 45 subjects is planned to achieve approximately 36 participants completing the study.

DETAILED DESCRIPTION:
After up to a 4-week screening period, participants will undergo 8 weeks of active or placebo treatment (Period 1), followed by an 8-week washout period, and then cross over to 8 weeks of placebo or active treatment (Period 2). Patients will be followed for 2 weeks after completion of Period 2. Two dosing groups are designated as Group A, who are randomly assigned to active treatment with KZ101 in Period 1 and saline in Period 2, and Group B, who are randomly assigned to saline infusion in Period 1 and active treatment with KZ101 in Period 2. Dosing in both periods will consist of 2 IV infusions of either saline (placebo) or KZ101 (active treatment), given 4 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

- Subject must meet all of the following criteria to be enrolled in this study.

1. Male, aged 5-14 years
2. Clinical diagnosis of ASD by DSM-5 criteria
3. ADOS-2 ≥ 7 on the comparison score for Modules 2-4 (completed within the last 2 years).
4. CGI-S ≥ 4 for socialization specific symptoms of ASD
5. Leiter-3 non-verbal IQ > 70
6. Standard score < 75 on the Socialization Domain of the Comprehensive Interview Form of the Vineland Adaptive Behavior Scale Third Edition
7. Subjects who are sexually active or potentially sexually active agree to use condoms with a spermicidal as a barrier method of contraception during the treatment period and for at least 30 days after the last dose of study medication
8. Subjects agree to wear sunscreen and to wear skin covering to the maximal degree tolerated by the child for the duration of the treatment period and for at least 30 days after the last dose of study medication
9. Subjects must have a ≤ 90 minutes car ride from the study site
10. English-speaking child and parent/guardian or caregiver
11. Parent or their legal guardians must be willing to sign informed consent

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from the study.

  1. ASD diagnosis with underlying syndromic diagnosis (e.g., Fragile X, Angelman, Down's Syndrome, etc.)
  2. ≤ 5th percentile for weight
  3. Unable to tolerate venipuncture or urine collection
  4. Acute infection (e.g., upper respiratory tract infection, common cold, flu, strep, COVID-19)
  5. Severe co-morbid conditions (e.g., psychosis, seizures/epilepsy uncontrolled by medication, presence of severe visual or hearing impairment) that may interact with study procedures. Controlled epilepsy is allowed providing there has not been a breakthrough seizure in the past year.
  6. Any organ system dysfunction, especially liver (e.g., ALT or AST ≥ 1.5x the upper limit of normal), kidney (estimated glomerular filtration rate or eGFR < 90 mL/min/1.73 m2; hematuria confirmed by urine microscopy [ > 5 red blood cells/high power field]; proteinuria [> 1+ that does not resolve on repeat testing or urine protein to creatinine ratio > 0.3]; and/or presence of any granular, mixed cellular, red blood cell, white blood cell, or muddy brown casts on urine microscopy), or clinically relevant heart or adrenal abnormalities
  7. Hospitalization within the previous 2 months from screening
  8. Initiation or change in pharmacotherapy within previous 2 months from screening
  9. Initiation or change in psychosocial interventions (formal behavioral, cognitive, or cognitive-behavior therapy) within previous 2 months from screening
  10. Plan to initiate or change pharmacotherapy or psychosocial interventions during the study
  11. Taking prescription medication that may interact adversely with KZ101 or expose the subject to increased risk of harm such as medications with plasma bound substances including sulfonamides, chlorpromazine, and anti-coagulants
  12. Currently enrolled in another clinical study or has received any investigational treatment within 30 days of screening
  13. Taking > 3 medications addressing behavioral symptoms related to ASD (ie typical/atypical antipsychotics and alpha-adrenergic agonists) or comorbid medical conditions such as ADHD, anxiety, or depression. Anti-seizure medications and other medications not related to neurobehavioral symptoms do not count towards the total number of medications allowed.
  14. History of serious dermatological reactions
  15. History of allergy, intolerance, or photosensitivity to any drug
  16. Unable or unwilling to adhere to study requirements

Ages: 5 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint - Vineland-3 Socialization Domain | Change from Screening to Week 8 (before washout) will be compared to change from Week 16 to Week 24 (after washout).
  The primary efficacy endpoint will be the change in standard score on the Socialization Domain of the Comprehensive Interview Form of the Vineland Adaptive Behavior Scale Third Edition (Vineland-3), which includes subdomains for coping skills, play skills, and interpersonal relation skills.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint - Vineland-3, Additional Scores | Secondary outcome measures will be used to assess change from Week 0 to Week 8 (before washout) and from Week 16 to Week 24 (after washout).
  Vineland-3 Composite Score, Communication Domain Score, and Daily Living Skills Domain Score will also be assessed.
Secondary Efficacy Endpoint - Global Impresssion, Severity/Change | Secondary outcome measures will be used to assess change from Week 0 to Week 8 (before washout) and from Week 16 to Week 24 (after washout).
  Clinician Global Impression of Severity and Change, and Caregiver/Parent Global Impression of Severity and Change, will be collected and assessed weighted for socialization.
Secondary Efficacy Endpoint - Social Responsiveness Scale-2 | Secondary outcome measures will be used to assess change from Week 0 to Week 8 (before washout) and from Week 16 to Week 24 (after washout).
  The Social Responsiveness Scale-2 (SRS-2) is a well-established tool to evaluate socialization that was also used in a prior pilot study.
Secondary Efficacy Endpoint - Aberrant Behavior Checklist, Second Edition (ABC-2) | Secondary outcome measures will be used to assess change from Week 0 to Week 8 (before washout) and from Week 16 to Week 24 (after washout).
  The ABC-2 provides measures of repetitive behaviors and includes domains of irritability, social withdrawal, stereotypy, hyperactivity, and inappropriate speech.
Secondary Efficacy Endpoint - Childhood Sleep Habits Questionnaire (CSHQ) | Secondary outcome measures will be used to assess change from Week 0 to Week 8 (before washout) and from Week 16 to Week 24 (after washout).
  As a large proportion of the adolescents with ASD population is highly impacted by sleep concerns, the CSHQ will be administered to investigate relationships between KZ101 and sleep.
Secondary Efficacy Endpoint - Parenting Stress Impact (PSI) | Secondary outcome measures will be used to assess change from Week 0 to Week 8 (before washout) and from Week 16 to Week 24 (after washout).
  Data from the PSI will be used to evaluate whether changes in symptoms in the ASD participant is associated with changes in parental stress throughout the study.
Secondary Efficacy Endpoint - Child Behavior Check List (CBCL) | Secondary outcome measures will be used to assess change from Week 0 to Week 8 (before washout) and from Week 16 to Week 24 (after washout).
  The CBCL is a parental measure of internalizing and externalizing behaviors as well as common DSM-5 conditions co-occurring with ASD.
Secondary Efficacy Endpoint - Ohio State University Autism Rating Scale, 5th Edition | Secondary outcome measures will be used to assess change from Week 0 to Week 8 (before washout) and from Week 16 to Week 24 (after washout).
  The Ohio State University Autism Rating Scale 5 (OARS-5) will provide three summary scores to be evaluated with KZ101 administration and placebo administration: autism symptom count, weighted mean severity score of autism symptoms, and impairment index based on level of support needed.

OTHER OUTCOMES:
Pharmacokinetic (PK) Endpoints: Cmax | PK samples will be taken at week 0, 2, 4, 6, 8 (period 1); and 16, 18, 20, 22, 24, 26 (period 2 and follow up).
  Blood samples for measurement of KZ101 concentration in plasma will be collected and used to identify Peak Plasma Concentration (Cmax).
Pharmacokinetic (PK) Endpoints: Area Under the Curve (AUC) | PK samples will be taken at week 0, 2, 4, 6, 8 (period 1); and 16, 18, 20, 22, 24, 26 (period 2 and follow up).
  Blood samples for measurement of KZ101 concentration in plasma will be collected, and area under the plasma concentration versus time curve (AUC) will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Aram Kim, MD, Principal Investigator — Thompson Autism and Neurodevelopmental Center, Children's Hospital of Orange County
Locations (3):
- United States (3):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Children's Hospital Orange County, Thompson Autism and Neurodevelopmental Center, Orange, California
  - Kennedy Krieger Institute, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.

REFERENCES:
- [Background] Naviaux RK, Zolkipli Z, Wang L, Nakayama T, Naviaux JC, Le TP, Schuchbauer MA, Rogac M, Tang Q, Dugan LL, Powell SB. Antipurinergic therapy corrects the autism-like features in the poly(IC) mouse model. PLoS One. 2013;8(3):e57380. doi: 10.1371/journal.pone.0057380. Epub 2013 Mar 13. PMID 23516405
- [Background] Naviaux JC, Schuchbauer MA, Li K, Wang L, Risbrough VB, Powell SB, Naviaux RK. Reversal of autism-like behaviors and metabolism in adult mice with single-dose antipurinergic therapy. Transl Psychiatry. 2014 Jun 17;4(6):e400. doi: 10.1038/tp.2014.33. PMID 24937094
- [Background] Naviaux JC, Wang L, Li K, Bright AT, Alaynick WA, Williams KR, Powell SB, Naviaux RK. Antipurinergic therapy corrects the autism-like features in the Fragile X (Fmr1 knockout) mouse model. Mol Autism. 2015 Jan 13;6:1. doi: 10.1186/2040-2392-6-1. eCollection 2015. PMID 25705365
- [Background] Naviaux RK, Curtis B, Li K, Naviaux JC, Bright AT, Reiner GE, Westerfield M, Goh S, Alaynick WA, Wang L, Capparelli EV, Adams C, Sun J, Jain S, He F, Arellano DA, Mash LE, Chukoskie L, Lincoln A, Townsend J. Low-dose suramin in autism spectrum disorder: a small, phase I/II, randomized clinical trial. Ann Clin Transl Neurol. 2017 May 26;4(7):491-505. doi: 10.1002/acn3.424. eCollection 2017 Jul. PMID 28695149
- See also: Thompson Autism and Neurodevelopmental Center, Clinical Trials — https://choc.org/research/autism-research/